CLINICAL TRIAL: NCT03753568
Title: Effect of an Electronic Reminder System on Direct Oral Anticoagulant and Oral Diabetes Medication Adherence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Janne Sahlman, Chief medical officer, Popit Ltd, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2018-11-21; First posted 2018-11-27 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Anticoagulant Drugs; Diabetes Mellitus, Type 2
Keywords: medicine reminder; diabetes mellitus, type 2; direct oral anticoagulants
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Subjects are monitored first before the intervention and then during the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): The participants use either direct oral anticoagulants or oral diabetic medication.
  Interventions: Device: Electronic medicine reminder system

INTERVENTIONS:
Device: Electronic medicine reminder system — Electronic surveillance device is attached to the participants push through pill sheet and the smart phone application reminds the participants to take their medicine if they are about to take their daily dosage.

SUMMARY:
In this study, the effect of an electronic device attached to a push through pill package and a smart phone application on chronic disease medication adherence is studied.

DETAILED DESCRIPTION:
In this study study two different groups of medicine users are recruited. Both groups have 50 patients each. In the first study the participants are using oral medication for diabetes and in the second study the participants use new direct oral anticoagulants.

Participants use medicine reminder system consisting of an electronic device and an smart phone application. In the beginning of the study the reminder system is collecting data on how the patients are taking their medication for the first two months. Smart phone application is not providing any reminders and participants can't access the app to see the details.

After two months the application will be unlocked so that it starts reminding the users to take their medication at the right time. in this phase the patients can view their medication data from the application. The reminder phase of the study lasts for two months. After these two plus two months, the results are analyzed and published.

The study continues after these four months for the next four months and after that, the long term results are analyzed.'

The primary outcome is the possible change in the adherence between control and active period.

ELIGIBILITY:
Inclusion Criteria:

* use of direct oral anticoagulants or oral diabetic drugs
* age of 18 or more
* subjects have been using a smart phone

Exclusion Criteria:

* patients who don't use their medication without help

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to the medication | 8 months
  PDC - proportion of days covered

SECONDARY OUTCOMES:
Variation of daily pill taking times | 8 months
  The mean difference from the mean pill taking time

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided